CLINICAL TRIAL: NCT01330849
Title: A Randomized Controlled Trial of a Behavior Modification Toolkit in Primary School Children With ADHD Behaviors
Brief Title: Toolkit for School Behavior Modification in Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Prof. dr. Marina Danckaerts, Universitaire Ziekenhuizen Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S52891
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-04

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; School; Behavioral Intervention; RCT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toolkit intervention (Experimental)
  Interventions: Behavioral: ADHD Toolkit
- Waiting List Control Group (No Intervention): Children eligible for the study according to the inclusion criteria, but randomly allocated to the waiting list control group are promised to receive the intervention AFTER the study is finished.
  Interventions: Other: Waiting List Control group

INTERVENTIONS:
Behavioral: ADHD Toolkit — For children allocated to the active intervention arm, teachers are trained to apply the ADHD Toolkit. Teacher will use the behaviour modification tool for 3 months. They are trained to select target behaviours causing impairment for the child and will apply a systematic approach of increased intensity of monitoring and feedback for the behaviour, including training of appropriate behaviour.
  Arms: Toolkit intervention
Other: Waiting List Control group — Children in the control group will receive no specific intervention, but are promised that their teachers will apply the schoolkit for them after the study.
  Arms: Waiting List Control Group

SUMMARY:
The purpose of this study is to examine the efficacy of the ADHD-Toolkit (a toolkit for school behaviour modification in primary school children with ADHD-behaviours) in terms of general improvement in ADHD symptoms, specific targeted school-related problem behaviours, other disruptive behaviour disorder symptoms, teacher attitudes towards ADHD, teacher-child relationship and child self-esteem.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a debilitating and common disorder of childhood marked by pervasive and persistent patterns of inattention, overactivity and impulsiveness. It is associated with impairment in a range of domains at both home and school and leads to long term educational and vocational underachievement, delinquency and conduct disorder and social and marital problems. Current treatment approaches involve both pharmacological and non-pharmacological options. Non-pharmacological options tend to focus on home-based approaches such as parent training. These can be effective especially in limiting impairment and reducing symptoms of comorbid problems such as oppositional defiant disorder (ODD) and other psychiatric comorbidities. This can really improve the quality of life of children with ADHD. However, a major problem with these home-based approaches is that their effects are unlikely to generalise to the school setting. This means that to effectively treat ADHD and to deal with impairment at both home and at school one needs to supplement home based approaches with effective school based strategies.

Classroom-based approaches that have been tried with ADHD can be divided into two types (Pelham & Fabiano, 2008). First, there are classroom based management strategies where teachers manipulate the consequences of behaviour to reduce (i.e., negatively reinforce) inappropriate behaviours (aggression, loss of concentration, disruptiveness) and increase (reinforce) appropriate behaviours (compliance, concentration). The second type of intervention focuses on academic targets through manipulating the academic instruction and materials (i.e., reducing task length, peer tutoring). In the current proposal the investigators focus on the first category. Pelham & Fabiano (2008) recently concluded that "the evidence for BCM [behavioural classroom management] for ADHD was substantial".

However, while there is a considerable evidence base for the value of classroom management as a component of ADHD treatment in multi-modal psychosocial treatment packages in school-aged children, there is a lack of well designed randomized studies in a naturalistic school setting that can provide a definitive estimate of efficacy for such approaches.

At the University Hospital of Leuven a toolkit for school behaviour modification in children with ADHD has been developed and piloted. This is an instrument for teachers to systematically target specific behaviours in the classroom and the playground with the ultimate goal of improving school ADHD behaviours and reducing oppositionality. Teachers will identify the behaviours which are most challenging and apply a series of levels of intervention with increasing intensity of monitoring, feedback and training. The effect of a three month application of the toolkit will be evaluated compared to a waiting list control group. Outcome measures will include measures of ADHD behaviours, oppositional defiant behaviour, teacher attitudes towards ADHD, teacher-child relationship and child self-esteem.

ELIGIBILITY:
Inclusion Criteria:

* The teacher must rate the ADHD symptoms of the student above or equal to the 90,9th percentile on the inattention or hyperactivity/impulsivity subscale of the VvGK (a Dutch translation of the Disruptive Behaviour Disorders Rating Scale).
* There is a maximum of 2 children per classroom that may be included.

Exclusion Criteria:

* None (Medication use would not be a reason for exclusion from the sample if children still fulfill the inclusion criteria)(Children with mental retardation (IQ < 70) will automatically be excluded from the study, since the study runs in normal schools.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
DBD Rating Scale: ADHD subscale, teacher rated | Evaluation after using the ADHD Toolkit for a three month period
  DBD = Disruptive Behaviour Disorder Rating Scale (Pelham et al, 1992), teacher rated.

SECONDARY OUTCOMES:
DBD Rating Scale: ADHD subscale, parent rated | Evaluation after using the ADHD Toolkit for a three month period
  DBD = Disruptive Behaviour Disorder Rating Scale (Pelham et al, 1992), parent rated
DBD Rating Scale, oppositional defiant disorder subscale, teacher rated | Evaluation after using the ADHD Toolkit for a three month period
  DBD = Disruptive Behaviour Disorder Rating Scale (Pelham et al, 1992), teacher rated
DBD Rating Scale, oppositional defiant disorder subscale, parent rated | Evaluation after using the ADHD Toolkit for a three month period
  DBD = Disruptive Behaviour Disorder Rating Scale (Pelham et al, 1992), parent rated
Target Behaviour Improvement Rating Scale, teacher rated | Evaluation after using the ADHD Toolkit for a three month period
  Target Behaviour Improvement Rating Scale = a 24-item questionnaire (unpublished) based on the 24 target school behaviours listed in the treatment manual of the ADHD Toolkit (URL: http://www.uzleuven.be/adhd-toolkit), each item is scored on a four-point Likert scale, teacher rated
TRF, subscale internalizing problems | Evaluation after using the ADHD Toolkit for a three month period
  TRF = Teacher Report Form (Achenbach, 1991)
CBCL, subscale internalizing problems | Evaluation after using the ADHD Toolkit for a three month period
  CBCL= Child Behavior Checklist (Achenbach, 1991)
IRS, teacher rated | Evaluation after using the ADHD Toolkit for a three month period
  IRS= Impairment Rating Scale (Fabiano et al, 2006), teacher rated
IRS, parent rated | Evaluation after using the ADHD Toolkit for a three month period
  IRS= Impairment Rating Scale (Fabiano et al, 2006), parent rated
Perceived Competence Scale for Children | Evaluation after using the ADHD Toolkit for a three month period
  Perceived Competence Scale for Children (Harter, 1985)
Student-Teacher Relationship Scale | Evaluation after using the ADHD Toolkit for a three month period
  Student-Teacher Relationship Scale (Pianta, 1991)
Teachers Beliefs and Attitudes towards ADHD Scale, teacher rated | Evaluation after using the ADHD Toolkit for a three month period
  Teachers Beliefs and Attitudes towards ADHD Scale = A 20-item questionnaire (unpublished) looking at attributions of cause of ADHD, characteristics of children with ADHD and treatment options for ADHD. This questionnaire is a modification of Charlotte Johnstons ADHD Beliefs and Attitudes Scale [Johnston, C.(2001). ADHD Beliefs and Attitudes Scale. Unpublished scale.]. Scoring on a seven-point Likert scale, teacher rated.
Feasibility, Acceptability and Usefulness Scale, teacher rated | Evaluation after using the ADHD Toolkit for a three month period
  Feasibility, Acceptability and Usefulness Scale = A 15-item questionnaire measuring the feasibility, acceptability and usefulness of the ADHD Toolkit intervention, scoring on a five-point Likert scale, teacher rated. This questionnaire was developed specifically for this study (unpublished).
Feasibility, Acceptability and Usefulness Scale, student rated | Evaluation after using the ADHD Toolkit for a three month period
  Feasibility, Acceptability and Usefulness Scale = An 11-item questionnaire measuring the feasibility, acceptability and usefulness of the ADHD Toolkit intervention, scoring on a five-point Likert scale, student rated. This questionnaire was developed specifically for this study (unpublished).
DBD Rating Scale, conduct disorder subscale, teacher rated | Evaluation after using the ADHD Toolkit for a three month period
  DBD = Disruptive Behaviour Disorder Rating Scale (Pelham et al, 1992), teacher rated
DBD Rating Scale, conduct disorder subscale, parent rated | Evaluation after using the ADHD Toolkit for a three month period
  DBD = Disruptive Behaviour Disorder Rating Scale (Pelham et al, 1992), parent rated

CONTACTS AND LOCATIONS:
Overall Officials: Marina Danckaerts, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitair Ziekenhuis Leuven, Leuven, Vlaams-Brabant, Belgium